CLINICAL TRIAL: NCT03888846
Title: Clinical Protocol for Administration of Topical Pentoxifylline Gel on Behcet's Disease Oral Ulcers
Brief Title: Topical Pentoxifylline Gel on Behcet's Disease Oral Ulcers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ipekyolu Ilac Ltd. Sti (Industry)
Collaborators: Istanbul University - Cerrahpasa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P104375V04
Record Dates: First submitted 2019-03-21; First posted 2019-03-25 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-08

CONDITIONS: Behçet Disease Affecting Oral Mucosa
MeSH Terms: interventions — Pentoxifylline; Colchicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Colchicine (Other): Colchicine therapy as part of supportive care routinely offered in Behcet's Clinic-Istanbul
  Interventions: Drug: Colchicine
- Topical Pentoxifylline Gel and Colchicine (Experimental): Topical Pentoxifylline Gel administration in addition to the colchicine therapy as part of supportive care routinely offered in Behcet's Clinic-Istanbul
  Interventions: Drug: Pentoxifylline; Drug: Colchicine

INTERVENTIONS:
Drug: Pentoxifylline — Topical gel version of pentoxifylline to be administered intraorally.
  Other Names: Trental
  Arms: Topical Pentoxifylline Gel and Colchicine
Drug: Colchicine — Colchicine therapy is provided to patients with oral ulcers as part of supportive care routinely offered by Behcet's Clinic-Istanbul.
  Other Names: Colchicum-Dispert

SUMMARY:
Although Behçet's Disease (BD) has no FDA-approved therapies, numerous clinical reports suggest that oral ulcers of BD may resolve when treated with systemic ingested pentoxifylline (PTX). The investigators here propose to investigate the therapeutic potential of PTX dissolved in muco-adherent formulation and directly applied to the oral lesions. This 60 patient proof of concept trial is designed to meet regulatory requirements for safety concerns while at the same time exploring the potential efficacy and clinical utility of this product. The investigators hypothesize that application of topical PTX will accelerate the healing of these lesions in a clinically meaningful way, and further hypothesize that topical PTX can become a valuable adjunct to any other systemic therapy for BD.

DETAILED DESCRIPTION:
Behçet's Clinic at Cerrahpaşa Medical Faculty at the University of Istanbul has a long history of supportive care for BD patients and is recognized as the world leader in this regard. According to the EULAR 2018 recommended guidelines of Behcet's Disease, the first line of therapy recommended against recurring oral ulcers is colchicine. However, a significant portion of the participants undergoing colchicine therapy does not have sufficient response and require subsequent immune modulatory therapy. By comparing participants receiving colchicine as part of supportive care to those who also receive topical pentoxifylline (PTX), the investigators seek to prove the concept that topical PTX may have clinical value. Additionally, the investigators seek to demonstrate the safety and practicality of using topical PTX in BD patients. If the PTX gel therapy provides a sufficient response in participants, these participants might not need to undergo immune modulatory therapies. The risks of PTX are well characterized and previously reported adverse events were primarily gastrointestinal. The investigators expect fewer GI symptoms to result from the topical PTX application. The investigators anticipate the benefits of PTX can be optimized by a topical application, but require a trial to test that hypothesis.

ELIGIBILITY:
Inclusion Criteria:

* Meets the International Study Group criteria for Behcet's Disease
* Presents with at least one active lesions accessible to measurement, the largest of which is to be designated as the index ulcer
* Index oral ulcer to be assessed should be in the easily accessible areas of the oral mucosa, and the oral ulcer first began within 48 hrs prior to enrollment
* Adult (>18 years) male or a non-pregnant, non-lactating female
* Has signed an Ethics Committee (EC) approved subject consent form
* Has completed all screening procedures satisfactorily, is deemed to be an acceptable subject and is otherwise eligible for entry into the study
* Is willing and able to comply with the protocol
* Is being treated with colchicine

Exclusion Criteria:

* Has a severe, acute, or chronic systemic disease other than Behcet's Disease such as congestive heart failure, hepatic failure, renal failure, systemic lupus erythematosus, Stevens-Johnson syndrome, ulcerative colitis, cancer, leukemia, diabetes, AIDS, or any other condition that is severely compromising the immune system
* Has received pentoxifylline in any form over the previous 60 days prior to enrollment
* Has experienced recent cerebral and/or retinal hemorrhage or in patients who have previously exhibited intolerance to pentoxifylline or methylxanthines such as caffeine, theophylline, and theobromine
* Has concomitant administration of strong CYP1A2 inhibitors (including e.g. ciprofloxacin or fluvoxamine) and other drugs that may increase the exposure to pentoxifylline
* Is receiving immune suppressing or modulating therapy (e.g., apremilast) or topical corticosteroids within 2 weeks prior to enrollment
* Is not being treated with colchicine
* Is under active treatment for dental conditions, such that multiple dental office visits would be required during the study period, or presents with oral conditions which are not thought to be related to Behcet's Disease and in the judgment of a qualified dentist, will require treatment during the study period
* Is suffering from any medical condition other than Behcet's Disease known to cause oral ulcerations, such as erosive lichen planus, benign mucous membrane pemphigoid, Systemic Lupus Erythematous, Crohn's disease, Reiter's syndrome, or AIDS. Has an eating disorder and/or psychiatric illness requiring treatment. Has a history of, or is currently exhibiting, any disease or condition, which, in the opinion of the principal investigator, would place the subject at increased risk during study therapy. Has any abnormality in hematological or biochemical variable, which, in the opinion of the principal investigator, would place the subject at increased risk during study therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2019-03-25 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Mean change in the speed of healing of the index oral ulcer | The participants will be assessed at seven time points starting at enrollment when the index ulcer is assigned until the complete healing(disappearance) of the index oral ulcer. This time frame is estimated to take two weeks (please see SoA in protocol).
  The size of the index oral ulcer will be measured at study enrollment and during the two week trial at seven time points (Please see Schedule of Activities in the protocol for more detail). The change in the size of the index ulcer will be compared between two study arms.
Mean change in the total number of oral ulcers | The participants will be assessed at seven time points starting at the enrollment visit until the end of study visit. This time frame is estimated to take two weeks.
  The total number of oral ulcer will be measured at study enrollment and during the two week trial at seven time points (Please see Schedule of Activities in the protocol for more detail). The total number of oral ulcers will be compared between two study arms.
Mean change in patient reported outcome pain scores | The participants will be assessed at sixteen time points starting at the enrollment visit until the final follow up visit.This time frame is estimated to take 45 days. Please see Schedule of Activities(SoA) in the protocol.
  Pain scores will be compared between two study arms as measuring pain offers an opportunity to correlate simple measurements of oral mucosal disruption with patient's fundamental disease experience.

SECONDARY OUTCOMES:
Behcet's Disease-Quality of Life Assessment Questionnaire | The participants will be assessed at eight time points starting at the enrollment visit until the final follow up visit.This time frame is estimated to take 45 days. Please see Schedule of Activities(SoA) in the protocol.
  Participant's quality of life will be assessed by a Behcet's Disease specific questionnaire prepared by key opinion leaders in the field of Behcet's Disease research at the University of Leeds. Please see the "Behcet's Disease Quality of Life Measure" in the appendix of the protocol for more details.
Behcet's Disease Activity Index | The participants will be assessed at eight time points starting at the enrollment visit until the final follow up visit.This time frame is estimated to take 45 days. Please see Schedule of Activities(SoA) in the protocol.
  Behcet's Disease Activity Index is prepared by International Society for Behcet's Disease to guide the doctor in assessing the disease activity.

CONTACTS AND LOCATIONS:
Overall Officials: Gulen Hatemi, MD, Principal Investigator — Istanbul Universitesi-Cerrahpasa
Locations (1):
- Istanbul Universitesi-Cerrahpaşa Tıp Fakültesi, İç Hastalıkları Anabilim Dalı-Romatoloji, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification will be available to other researchers.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Beginning 3 months following publication. No end date.
Access Criteria: Proposals should be directed to bderkunt@gmail.com. Anyone who provides a methodologically sound proposal will be approved to perform any type of analysis to achieve the aims in the proposals. To gain access, data requestors will need to sign a data access agreement. Data will be made available indefinitely at (link to be included).

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-21): https://cdn.clinicaltrials.gov/large-docs/46/NCT03888846/Prot_SAP_000.pdf